CLINICAL TRIAL: NCT02625077
Title: Valvuloplasty as Alternative to Toupet Fundoplication for the Minimal Invasive Treatment of Gastroesophageal Reflux Disease: A Randomized Controlled Trial
Brief Title: Valvuloplasty as Alternative to Toupet Fundoplication for GERD
Acronym: VANTAGE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Ethical concerns with efficacy of technique.
Sponsor: Meander Medical Center (Other)
Responsible Party: Principal Investigator, R.C. Tolboom, MD, Project Leader, Meander Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHI-UPPERGI-VANTAGE; NL52398.100.15 (Registry Identifier: CCMO Register)
Record Dates: First submitted 2015-11-15; First posted 2015-12-09 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Gastroesophageal Reflux; Hernia, Hiatal
Keywords: Valvuloplasty; Fundoplication; Acid reflux; GERD; Reflux disease; Hiatal hernia
MeSH Terms: conditions — Gastroesophageal Reflux; Hernia, Hiatal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic valvuloplasty (Experimental): Via laparoscopy, using three sutures a part of the esophagus is folded (similar to the way parts of a telescope slide in each other) into the stomach, creating a valve on the inside to prevent gastric acid to enter the esophagus.
  Interventions: Procedure: Laparoscopic gastroesophageal valvuloplasty
- Laparoscopic Toupet fundoplication (Active Comparator): Via laparoscopy, the entire stomach is mobilized and folded around itself posteriorly, creating a partial (270 degrees) fundoplication.
  Interventions: Procedure: Laparoscopic Toupet fundoplication

INTERVENTIONS:
Procedure: Laparoscopic gastroesophageal valvuloplasty
  Arms: Laparoscopic valvuloplasty
Procedure: Laparoscopic Toupet fundoplication
  Arms: Laparoscopic Toupet fundoplication

SUMMARY:
This monocenter randomized controlled trial aims to compare postoperative outcomes of a laparoscopic valvuloplasty with a Toupet fundoplication in patients with GERD with a maximum hiatal hernia of 3cm. In addition, an economic evaluation of the new intervention will be done in order to determine cost-effectiveness and costs per quality-adjusted life-year (QALY).

DETAILED DESCRIPTION:
This is a prospective, interventional, double-blinded, monocenter randomized controlled trial comparing a laparoscopic gastroesophageal valvuloplasty to laparoscopic Toupet fundoplication in patients with proven GERD with a maximum hiatal hernia of 3cm. In this design, both patient and researcher are blinded to the treatment allocation.

Block randomization will be used to ensure an equal number in each treatment arm. Block randomization works by randomizing participants within blocks such that an equal number are assigned to each treatment. To reduce selection bias by predictability of the treatment allocation, random block sizes are used. Also the investigator is kept blind to the size of each block. A computer is used to generate 15 blocks for each participating center with random block sizes of 4, 8 and 12. Allocation proceeds by randomly selecting one of the orderings and assigning the next block of participants to study groups according to the specified sequence.

Patients will be included during a two-year period and followed for a minimum of one year. When a patient is referred to a participating surgeon for antireflux surgery, he or she will receive study information to give them sufficient time for consideration. The surgeon will ensure all required pre-operative diagnostic tests are performed and that the indication for surgery is valid. During a follow-up visit, the surgeon ascertains that the patient complies with all inclusion criteria and does not meet any of the exclusion criteria. Study participation will be discussed and after informed consent is obtained, the patient will be included in the trial.

After inclusion, the patient is immediately randomized but treatment allocation is not yet shared with the surgeon. The patient will receive validated questionnaires to record the pattern of symptoms, quality of life, medication and medical care usage. Data from the pre-operative tests will be recorded.

On the day of surgery, the surgeon will be able to see treatment allocation and after performing the appropriate surgical procedure, records the course and specifics of the surgical procedure. Patients will receive a diary to record their meals and symptoms.

Follow-up in the outpatient clinic will take place at the surgeon's discretion. At fixed moments: 3, 6 and 12 months after surgery, the patients will once more receive validated questionnaires. Also at about three months, a follow-up manometry and 24-hour pH and/or impedance monitoring will be performed.

A power analysis was performed to calculate the sample size. Our primary aim was to compare the effect of both surgical procedures. Based upon the current medical literature, the objective/subjective success rate for the laparoscopic Toupet fundoplication is around 88%. Pilot data from a retrospective cohort of patients that underwent valvuloplasty report a subjective success rate of 96%. Our hypothesis was that the gastroesophageal valvuloplasty is not inferior to the Toupet fundoplication when comparing its effects on acid control.

To prove non-inferiority of the valvuloplasty regarding acid reflux control, using a non-inferiority limit of 5%, 73 patients are required in each group. In all power calculations, a significance of 5% and power of 90% was used.

To accommodate for a loss to follow-up of up to 10 percent, a total sample size of 160 was chosen.

ELIGIBILITY:
Inclusion Criteria:

* Objectively proven GERD (by gastroscopy and/or 24-hour pH and/or impedance monitoring)
* Age ≥18
* Written informed consent for study participation

Exclusion Criteria:

* BMI ≥ 30
* Hiatal hernia >3cm
* Achalasia
* Previous gastric surgery
* Previous esophageal surgery
* Inability to understand the Dutch language
* Inability to understand and/or fill in the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Success rate, objective | 3 months post-operative
  Defined as % of patients with normal values of reflux measured by pH and impedance monitoring

SECONDARY OUTCOMES:
Success rate, subjective | 3 months post-operative, 1 year post-operative
  Defined as % of patients with Visick score I or II
Percent of patients with complaints of functional dysphagia according to the Rome III criteria | 3 months post-operative, 1 year post-operative
  % of patients with complaints of functional dysphagia according to the Rome III criteria.
Cost-effectiveness | 1 year post-operative
  Cost-effectiveness will be calculated by comparing the direct and indirect medical cost related to both strategies up until one years after the operation.
Mortality rate | 30 days
  Defined as in-hospital mortality or out of hospital mortality within 30 days
Complication rate | During surgery
  Intra-operative complication rate
Conversion rate | During surgery
Disease related reoperation rate | 1 year
  % of patients requiring redo surgery for persisting complaints or recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Werner A Draaisma, MD, PhD, Study Director — Meander Medical Center; Ivo AM Broeders, MD, PhD, Principal Investigator — Meander Medical Center
Locations (1):
- Meander Medical Center, Amersfoort, Utrecht, Netherlands

REFERENCES:
- See also: Meander Medical Center — http://www.meandermc.nl